CLINICAL TRIAL: NCT04372355
Title: Effect of WF10 (TCDO) on HbA1c Values in Diabetic Foot Ulcer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Srinakharinwirot University (Other)
Collaborators: Oxo Chemie(Thailand) Co.,Ltd. (Unknown); Altermed Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Narongchai Yingsakmongkol, Associate Professor, Srinakharinwirot University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SWUEC-043/2019F; WF10-19-THAI-01 (Other: SWU Ethical Committee)
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Foot Ulcer (DFU); Uncontrolled Diabetes With Foot Ulcer
Keywords: DFU; WF10
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: T2DM patients with DFU and HbA1c > 8.5%
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chlorite-based drug WF10 (Experimental): WF10, the chlorite-based drug is infused at a dose of 0.3 ml/Kg BW, after dilution in 300 mL physiological saline, over a period of 3 h. The drug is applied once a week for five
  Interventions: Drug: WF10

INTERVENTIONS:
Drug: WF10 — WF10, the chlorite-based drug is infused at a dose of 0.3 ml/Kg BW, after dilution in 300 mL physiological saline, over a period of 3 h. The drug is applied once a week for five subsequent weeks.
  Other Names: Immunokine

SUMMARY:
Study in adult Diabetes Mellitus patients with diabetic foot ulcers and elevated HbA1c who will receive standard wound treatment in combination with adjuvant therapy WF10 to compare the change of HbA1c levels at baseline and after treatment.

DETAILED DESCRIPTION:
Single-center, Prospective Open-labelled One Group Pretest Posttest Pilot Study

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Diabetes Mellitus type II
* Patient male or female 18-80 years old
* Presence of Diabetic foot ulcer/non-healed stump, starting at least 3 weeks before or infected wound degree 3-4
* HbA1c > 8.5%
* Hematocrit > 30%

Exclusion Criteria:

* Kanofsky performance status < 60
* Patient with ABI (Ankle Brachial index) < 0.4
* Patient who receive steroid ,chemotherapeutic drug
* Pregnant or lactating woman
* Patient had a history of organ transplantation, and using immunosuppressive drug
* Patient with end-stage renal disease requiring hemodialysis, or history of G6PD or severe thalassemia, or ischemic heart disease, Congestive heart failure, Heart arrhythmia
* Patient who is participating in another clinical study or have done it in the past 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
HbA1c change at Week 8 in comparison to Baseline | 8 weeks
  The mean change of HbA1c values between Baseline (Week 0) and Week 8 after the initial WF10 treatment

SECONDARY OUTCOMES:
HbA1c change at Week 12 in comparison to Baseline | 12 weeks
  The mean change of HbA1c values between Baseline (Week 0) and Week 12 after the initial WF10 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Narongchai Yingsakmongkol, MD, FRCST, Principal Investigator — Srinakharinwirot University
Locations (1):
- HRH Princess Maha Chakri Sirindhorm Medical Center, Ongkharak, Changwat Nakhon Nayok, Thailand

IPD SHARING:
Plan to Share IPD: No